CLINICAL TRIAL: NCT05227352
Title: Exploring the Concepts of Bio-experiential Spaces
Brief Title: Bio-Experiential Spaces for Mental Health in Healthworkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, David Putrino, Professor Rehabilitation and Human Performance, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY-21-01221
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-09

CONDITIONS: Mental Health; Cognition; Anxiety
Keywords: biophilic design; mental health; cognition; PTSD; anxiety; stress
MeSH Terms: conditions — Psychological Well-Being; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Biophilic experience (Experimental): Healthcare workers will experience the biophilic-designed room
  Interventions: Behavioral: Biophilic design experience

INTERVENTIONS:
Behavioral: Biophilic design experience — Recharge Rooms are immersive, biophilic private spaces featuring multisensory input that is inspired by nature.

SUMMARY:
Recharge Rooms are immersive, biophilic private spaces designed to ameliorate trauma, anxiety, and stress. They feature multisensory input that is inspired by nature, as has previously been found to confer physiological benefits. These environments include silk imitation plants, projected scenes of soothing natural landscapes, low lighting that is tailored in color to match the landscapes that are being projected, high definition audio recordings of nature sounds paired with relaxing music, and infusion of essential oils and calming scents.

The aim is to investigate the physiological and mental health outcomes that the short and long term exposure to these rooms have on healthcare workers. The data will be collected through online surveys. No identifiable information will be assessed or collected. The plan is to have 60 participants.

ELIGIBILITY:
Inclusion Criteria

* Adults over the age of 18
* Current healthcare employee of Mount Sinai Hospital or the Icahn School of Medicine at Mount Sinai

Exclusion Criteria

* Age under 18
* Not employed by Mount Sinai or Icahn School of Medicine at Mount Sinai

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Well-Being Index | 6 weeks
  This assesses a variety of dimensions such as burnout, fatigue, mental and physical quality of life (QOL), depression and anxiety, and is used as a screening tool to assess residents at "high risk," who may be in distress, and who benefit from added resources and subsequent help seeking. It uses yes/no response categories, and a total score is calculated by adding the number of 'yes' responses. Full scale range from 0 to 7, with higher score indicating poorer health outcome, and a threshold score of 5 is used to identify "high risk" residents.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder 7 (GAD7) | 6 weeks
  This 7-item instrument uses some of the DSM-V criteria for GAD (General Anxiety Disorder) to identify probable cases of GAD along with measuring anxiety symptom severity. It can also be used as a screening measure of panic, social anxiety, and PTSD. Responders are asked to rate the frequency of anxiety symptoms in the last 2 weeks on a Likert scale ranging from 0-3. Items are summed to provide a total score. Full scale from 0-21, with higher score indicating more symptoms.
The Patient Health Questionnaire (PHQ-9) | 6 weeks
  This is the major depressive disorder (MDD) module of the full PHQ. It is one of the most validated tools in mental health and can be a powerful tool to assist clinicians with diagnosing depression and monitoring treatment response. It is not a screening tool for depression but it is used to monitor the severity of depression and response to treatment. The nine items of the PHQ-9 are based directly on the nine diagnostic criteria for major depressive disorder in the DSM-IV. It scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). Total scores of 5, 10, 15, and 20 represent cut points for mild, moderate, moderately severe and severe depression, respectively . Full scale from 0-27, with higher score indicating more severe symptoms.
The Insomnia Severity Index (ISI) | 6 weeks
  This is a brief instrument that was designed to assess the severity of both nighttime and daytime components of insomnia. There are seven questions and the total score is found by summing the answers to the seven questions. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28). The total score ranges from 0-28 where higher score indicates increased severity of insomnia.
The Fatigue Severity Scale (FSS) | 6 weeks
  This is a 9-item scale which measures severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. The items are scored on a 7 point scale with 1=strongly disagree and 7=strongly agree. Full scale from 9 - 63, with higher score indicating greater fatigue severity.
Brief Resilience Scale (BRS) | 6 weeks
  This is a self-rating questionnaire aimed at measuring an individuals' ability to "bounce back from stress". The possible full scale range on the BRS is from 1 (low resilience) to 5 (high resilience), with higher score indicating higher resilience. The scores can be interpreted as follows: 1.00-2.99= low resilience; 3.00-4.30= normal resilience; 4.31-5.00= high resilience.
Satisfaction With Life Scale (SWLS) | 6 weeks
  SWLS is designed to measure global cognitive judgments of satisfaction with one's life. The scale usually requires only about one minute of a respondent's time. Life satisfaction is one factor in the more general construct of subjective well-being. The SWLS is a 7-point Likert style response scale. The full scale range is from 5-35, with a higher score indicating higher levels of life satisfaction. A score of 20 representing a neutral point on the scale. Scores between 5-9 indicate the respondent is extremely dissatisfied with life, whereas scores between 31-35 indicate the respondent is extremely satisfied.
Maslach Burnout Inventory-Human Services Survey | 6 weeks
  This measures the degree of burnout. Within the survey 3 domains are evaluated: Emotional Exhaustion (EE), 9 questions; Depersonalization (DP), 5 questions; and Personal Accomplishment (PA), 8 questions. All MBI-HSS items are scored on a Likert scale ranging from "never"=0 to "daily"=6. Scores from within each domain are added up and participants are classified into tiers (High, Moderate or Low) per domain. A high score of EE (score of 27 or higher) or a high score of DP (total score of 10 or higher) is considered indicative of clinically significant burnout in medical trainees.
Social Connectedness Scale | 6 weeks
  This assesses the degree to which you feel connected to others in social environments.The is a 20-item questionnaire that scales responses from 1 (strongly disagree to 6 (strongly agree). The items are summed with full range scale from 20 - 120; a higher score indicates more connectedness to others.
Situational Awe Scale | 6 weeks
  This is a self-reported measure to assess the momentary phenomenological experience of awe. 30-item instrument, each item scored on a 7-point scale: -3 (disagree strongly) to +3 (agree strongly). Full scale from 30 - 210, higher score indicates a stronger experience of awe.
Heart Rate Pulse Oximeter | 6 weeks
  This will be used to noninvasively measure heart rate (HR). Pulse oximetry is used to measure the oxygen level of the blood by using infrared light. The device will be placed on the participant's finger. The normal range for resting heart rate is between 60-100 beats per minute.
Oxygen Saturation (pO2) Oximeter | 6 weeks
  This will be used to noninvasively measure oxygen saturation (pO2). Pulse oximetry is used to measure the oxygen level of the blood by using infrared light. The device will be placed on the participant's finger. The normal range for oxygen saturation is 89-100%.
Automatic Blood Pressure | 6 weeks
  This will be used to measure blood pressure. The normal level for systolic blood pressure is less than 120 mmHg. The normal level for diastolic blood pressure is less than 80 mmHg.
Galvanic Skin Response (GSR) | 6 weeks
  This is one of the most sensitive measures for emotional arousal. Galvanic Skin Response originates from the autonomic activation of sweat glands in the skin. The sweating on hands and feet is triggered by emotional stimulation: Whenever a person is emotionally aroused, the GSR data shows distinctive patterns that are visible with bare eyes and that can be quantified statistically. A GSR device containing two electrodes will be placed on the skin of the participant during the Recharge Room experience. GSR is measured in the unit of microSiemens. Measurements normal range: 0-15 microSiemens.
Power spectrum density by EEG | 6 weeks
  Quantitative electroencephalography (EEG) power spectrum density. Mean power is the percentage of change between PRE and POST of the average power along time in each frequency band and electrode.
Coherence by EEG | 6 weeks
  Quantitative electroencephalography (EEG) coherence. Mean coherence is the percentage of change between PRE and POST of the mean coherence in each band and each electrode, defined as the average coherence of this electrode with all the other ones.
Frequency band power by EEG | 6 weeks
  Quantitative electroencephalography (EEG) frequency band power. Mean frequency is the percentage of change between PRE and POST of the mean frequency in each band and electrode, defined as the mean frequency of the power spectrum weighted over that band.

CONTACTS AND LOCATIONS:
Overall Officials: Mar Cortes, MD, Principal Investigator — Icahn School of Medicine
Locations (1):
- Recharge Room at Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD at this time.

DOCUMENTS (1):
  • Informed Consent Form (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT05227352/ICF_000.pdf